CLINICAL TRIAL: NCT07172113
Title: Utilizing Embodied Artificial Intelligence (AI) for the Development of Digital Cognitive Behavioral Therapy (CBT) for Depression in Virtual Reality (VR): a Pilot RCT
Brief Title: Utilizing Embodied Artificial Intelligence (AI) for the Development of Digital Cognitive Behavioral Therapy (CBT) for Depression in Virtual Reality (VR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tim M. H. Li, Prof., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024.061
Record Dates: First submitted 2025-03-11; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Depression Scale Score

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The VR group will receive one session CBT via a VR headset. The session will last for around 45 mins. During the intervention, the participants can freely talk to the virtual therapist using natural language input.
  Interventions: Device: CBT + VR
- Control group (No Intervention): This group will serve as a waitlist control group. They will not receive the intervention until the study end.

INTERVENTIONS:
Device: CBT + VR — This CBT intervention is conducted in VR using Embodied AI technology. A virtual therapist will present in a virtual therapy room. Participants can freely talk to and interactive with the virtual therapist.
  Arms: Intervention group

SUMMARY:
Depression is a prevalent mental disorder characterized by pervasive low mood, diminished interest or pleasure, and a range of cognitive and physical symptoms. According to the World Health Organization (WHO), depression is a leading cause of disability worldwide, affecting approximately 280 million individuals of all ages. In spite of the widespread occurrence and negative consequences linked to depression, fewer than 30% of individuals with common mental disorders sought assistance from mental health services in the previous year due to reasons such as, high-cost and stigma.

Cognitive behavioral therapy (CBT) is the gold-standard and evidence-based intervention for various mental health disorders, including depression, anxiety, and its effectiveness has been widely proven. With the recent advancement in AI and other relevant technologies, the use of digital CBT has become possible. Indeed, a recent systematic review demonstrated a comparable effectiveness of traditional CBT and digital CBT, after controlling the moderators (e.g., intervention duration, and adherence). While digital CBT has achieved impressive performance, the majority of them utilized web-based or app-based platforms. Therefore, one of the disadvantages of such digital CBT is the lack of interaction between (digital) therapists and clients. Additionally, lower adherence to digital interventions was observed, indicating the need for briefer sessions, such as single-session integrated CBT (SSI-CBT), for digital interventions. SSI-CBT involves a collaborative effort between the therapist and the client, aimed at assisting the client in accomplishing their desired outcome within a single session. It is understood that additional support is accessible if required. A recent study using SSI-CBT demonstrated promising results of its effectiveness in reducing depression and anxiety, which can last for two months. To further generalize the application of digital interventions, a more interactive virtual therapist utilizing a brief CBT-based intervention approach is desired.

This study will evaluate the effectiveness of virtual CBT therapist for reducing depression symptoms, compared to a waitlist control group. Based on previous research, it is expected that a virtual CBT therapist can significantly reduce the depression symptoms at both post-intervention and one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese young adult aged 18-40 years
2. Native Cantonese speaker
3. Presence of depressive symptoms, as indicated by a score of 10 or higher on the depression sub-scale of the Depression Anxiety Stress Scale 21 (DASS-21).
4. Able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

1. A current or history of any psychiatric disorder(s) other than depressive disorder and anxiety disorder, such as bipolar disorder, psychotic disorders, and substance use disorder
2. A current or history of any voice, speech, and language disorders
3. A current or history of non-suicidal self-injury or suicidality
4. Incompetent in giving informed consent for participation in the study
5. A current or history of significant motion sickness, active nausea, and vomiting or epilepsy.
6. A current or history of color vision deficiency
7. Subject who is preparing for pregnancy or pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The Depression Subscale of the Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | Baseline and 1 month
  The depression sub-scale of DASS-21 comprises seven items that are assessed on a 4-point Likert scale, ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much). The international cut-off values are as follows (as multiplication of sum by 2): 0-9 for normal, 10- 13 for mild, 14- 20 for moderate, 21- 27 for severe and 28 or above for extremely severe.

SECONDARY OUTCOMES:
The Satisfaction With Life Scale (SWLS) | Baseline and 1 month
  The SWLS, containing 5 items, will be used to assess participants' life satisfaction. Items are scored based on a 7-point scale from strongly disagree (1) to strongly agree (7). A higher mean score indicates a greater satisfaction with life.
The revised General Help-Seeking Questionnaire (GHSQ) | Baseline and 1 month
  The revised GHSQ contained first 10 questions from the original GHSQ, asking people's intention to seek help from various sources, and further incorporated 9 follow-up questions, asking people's attitude to seek help from various sources. All items are scored based on a 7-point scale, ranging from extremely unlikely (1) to extremely likely (7) for the first 10 intention-related items, and from extremely unhelpful (1) to extremely helpful (7) for the last 9 attitude-related items. A higher mean score indicates a greater intention and attitude to seek help.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided